CLINICAL TRIAL: NCT00427414
Title: Pilot Study of Viral Load and Transcription in Kaposi's Sarcoma Patients Treated With Liposomal Anthracyclines
Brief Title: Liposomal Daunorubicin in Treating Patients With HIV-Related Kaposi's Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-050; U01CA070019 (NIH); CDR0000526564 (Other: NCI)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- liposomal daunorubicin citrate (Experimental): 40 mg/m2 Days 1 and 15 every 28 days x 3 cycles
  Interventions: Drug: liposomal daunorubicin citrate

INTERVENTIONS:
Drug: liposomal daunorubicin citrate — 40 mg/m2 Days 1 and 15 every 28 days x 3 cycles
  Other Names: DaunoXome

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal daunorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This clinical trial is studying how well liposomal daunorubicin works in treating patients with HIV-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of liposomal daunorubicin citrate on Kaposi's sarcoma-associated herpes virus (KSHV) viral gene expression in tumors of patients with HIV-related Kaposi's sarcoma.

Secondary

* Determine the effect of this drug on KSHV viral gene expression in peripheral blood mononuclear cells.
* Determine the effect of this drug on KSHV viral load in plasma.
* Correlate viral load with viral gene expression and/or tumor regression in these patients.

OUTLINE: This is a multicenter, pilot study.

Patients receive liposomal daunorubicin citrate IV days 1 and 15. Treatment repeats every 4 weeks for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Biopsies are performed at baseline and once during treatment to evaluate Kaposi's sarcoma- associated herpes virus (KSHV) viral gene expression in tumors and skin tissue using reverse transcriptase-quantitative polymerase chain reaction. Blood samples are collected at baseline and periodically during treatment to evaluate KSHV viral gene expression in peripheral blood mononuclear cells and viral load in plasma.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Kaposi's sarcoma (KS) involving the following:

  * Skin
  * Lymph nodes (palpable disease only)
  * Oral cavity
* Must have ≥ 5 measurable, previously nonirradiated, cutaneous lesions that can be used as indicator lesions
* Must have 2 lesions ≥ 5 x 5 mm that are accessible for 4 mm punch biopsy
* Serologically confirmed HIV positivity
* Concurrent antiretroviral therapy required, except for patients who have exhausted all available treatment options

  * Must be on a stable dose for ≥ 4 weeks

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* No other neoplasia requiring cytotoxic therapy
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior anthracycline therapy
* At least 4 weeks since prior antineoplastic treatment for KS, including any of the following:

  * Chemotherapy (6 weeks for nitrosoureas or mitomycin C)
  * Radiotherapy
  * Local therapy
  * Biological therapy
  * Investigational therapy
* At least 60 days since prior local therapy of any KS indicator lesion unless lesion has clearly progressed since treatment
* No other concurrent investigational drugs, cytotoxic chemotherapy, or KS-specific treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effect of liposomal daunorubicin citrate on Kaposi's sarcoma-associated herpes virus (KSHV) viral gene expression in tumors | 24-48 hours after the first treatment

SECONDARY OUTCOMES:
Effect of treatment on KSHV viral gene expression in peripheral blood mononuclear cells | 24-48 hours after treatment on Day 1/cycle 1, Day 8/cycle 1, and Day 29/cycle 3
Effect of treatment on KSHV viral load in plasma | 24-48 hours after treatment on Day 1/cycle 1, Day 8/cycle 1, and Day 29/cycle 3

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Ramos, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center; Dirk Dittmer, PhD, Study Chair — UNC Lineberger Comprehensive Cancer Center; Tamara Newman Lobato Souza, Principal Investigator — Instituto De Infectologia Emilio Ribas Hospital; Luis Carlos Pereira, MD, Principal Investigator — Instituto De Infectologia Emilio Ribas Hospital
Locations (3):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States
- Brazil (2):
  - Centro de Referencia e Tratamento DST/AIDS, São Paulo, São Paulo
  - Instituto De Infectologia Emilio Ribas Hospital, Cerqueira Cesar - Sao Paulo/SP